CLINICAL TRIAL: NCT01127867
Title: Docosahexaenoic Acid (DHA) Reduces Inflammation and Aromatase Expression in Subcutaneous Fat in Obese Postmenopausal Women: A Pilot Study
Brief Title: A Pilot Study of Docosahexaenoic Acid (DHA) in Obese Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PHO-0702
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer; Obesity
MeSH Terms: conditions — Breast Neoplasms; Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: dietary intervention — dietary intervention

SUMMARY:
This study aims to determine if a supplement of an omega-3-fatty acid (docosahexaenoic - DHA) lowers inflammation in human fat tissue thereby lowering estrogen production and the potential risk for breast cancer. The investigators also aim to study how this occurs to discover the basis for other potential treatments to lower estrogen production in fat tissue and decrease the risk of breast cancer.

DETAILED DESCRIPTION:
Breast cancer is one of the most frequently seen cancers in the United States. Breast cancer occurs at all ages but is particularly common in post menopausal women. Obesity increases the risk of breast cancer primarily of the type that is stimulated by the female sex hormone estrogen. In obesity, fat cells produce estrogen which can alter breast tissue, while lowering blood estrogen reduces the incidence of breast cancer. Inflammation of fat tissue, the coronary blood vessels and the liver are also seen with obesity. Animal experiments have shown the inflammation in fat tissue increases the production of estrogen, thus reducing inflammation in fat tissue might lower estrogen levels and the risk of breast cancer in obese women. A diet high in omega-3-fatty acids, such as those found in fish oil, has been shown in mice to reduce inflammation and aromatase expression (rate limiting enzyme for estrogen synthesis) in fat tissue.

This pilot study of five obese, post-menopausal women and an additional 12 morbidly obese post-menopausal women will include nutritional and medical evaluations, a four day inpatient hospital stay on a regular diet, to measure the inflammation and the estrogen producing machinery of each volunteer subject. Following these baseline measurements, subjects will be provided DHA supplements to take daily for three months and requested to weigh themselves twice weekly at home with the goal of maintaining their weight. Telephone interviews will be performed at scheduled points to check-in with the subjects and after six weeks a return visit to the OPRC will be conducted to assess progress and provide additional supplements. At three months each subject will be readmitted to the hospital and repeat the tests performed before starting on the DHA supplement. If the study shows feasibility and positive results it will be extended to more subjects and other interventions in the future.

ELIGIBILITY:
Inclusion Criteria:

Post-menopausal defined as:

1. 24 consecutive months without a menstrual period AND
2. low serum estradiol level (<40 ng/ml) to be assessed at screening AND
3. not taking any medication known to induce ammenorrhea AND
4. no known endocrine abnormality associated with irregular/absent menses.
5. BMI 35-50.

Exclusion Criteria:

1. Currently taking any hormone therapy: oral, transplanted, vaginal, injected
2. Currently taking NSAIDS (if > once a week, stopped < 30 days ago)
3. Currently taking oral hypoglycemics
4. Currently taking anticoagulant mediation or stopped < 30 days ago
5. History of any malignancy or cancer treatment in the past 3 years
6. Blood Pressure > 150/90 at screening
7. History of any bleeding disorder
8. Screening LFT results > 2x normal upper limits
9. Screening renal lab results > 2x normal upper limits
10. Any condition or situation which, in the investigator's opinion, puts the patient at significant risk, could complicate the study results, or may interfere significantly with participation in the study.
11. History of intestinal malabsorption
12. Screening urinalysis positive for blood
13. History of chronic diarrhea
14. History positive for HIV
15. Currently on any medication that can alter fat stores or large bowel inflammation as deemed by the principal investigator
16. History of inflammatory bowel disease
17. Screening thyroid function test abnormal
18. Currently taking any weight control medication
19. HIV positive as per POCT rapid test at screening
20. Currently taking fish oil, omega-3 supplements or other herbals that exceed the GRAS (Generally Recognized As Safe) levels
21. Fasting blood sugar greater than 126 mg/dL at screening
22. Currently taking more than 3 antihypertensive medications

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Reduced subcutaneous fat (obese) | 6 weeks
  Reduced subcutaneous fat inflammation changes between pre and post treatment for 5 pilot subject as seen by histologic quantification of monocyte aggregations (crowns), CD68 and CD163 stained macrophages in fat biopsies.
Reduced subcutaneous fat (morbidly obese) | 6 weeks
  Reduced subcutaneous fat between pre and post treatment for an additional 12 morbidly obese subjects as seen by histologic quantification of monocyte aggregations (crowns), CD68 and CD163 stained macrophages in fat biopsies.

SECONDARY OUTCOMES:
multiplex bead assay/immunoassay | 6 weeks
  Lowered aromatase expression in fat biopsies accompanied by decreases in the synthetic enzyme COX1-MPGES-1 and/or increase in the catabolic enzyme 15-PGDH and associated changes in BRAC-1 and SIRT-1 expression by immunohistochemical evaluation of CD68, CD168 and CD3 stained monocytes and through examination of the mRNA of imune inflammatory markers in fat biopsies.
  Alteration in serum estradiol and testosterone levels and/or changes in circulating cytokines/chemokines measured by multiplex bead assay and immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Holt, MD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The Rockefeller University clinical research information page — http://rucares.org